CLINICAL TRIAL: NCT05083182
Title: A Phase 3 Multicenter, Open-label Study to Evaluate the Efficacy, Pharmacokinetics, Safety, and Immunogenicity of Subcutaneously Administered Ustekinumab or Guselkumab in Pediatric Participants With Active Juvenile Psoriatic Arthritis (PSUMMIT-Jr)
Brief Title: A Study of Ustekinumab or Guselkumab in Pediatric Participants With Active Juvenile Psoriatic Arthritis
Acronym: PSUMMIT-Jr
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR109101; CNTO1275JPA3001 (Other: Janssen Research & Development, LLC); 2020-005503-40 (EudraCT Number)
Record Dates: First submitted 2021-10-08; First posted 2021-10-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Arthritis, Juvenile
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Ustekinumab; guselkumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Ustekinumab (Experimental): Participants will receive a weight-based dose of ustekinumab subcutaneously (SC) at Week 0, Week 4 and then every 12 weeks up to Week 52. Cohort 1 is closed for further enrollment.
  Interventions: Drug: Ustekinumab
- Cohort 2: Guselkumab (Experimental): The dose of guselkumab will be based on the participant's weight. Participants will receive guselkumab SC at Weeks 0 and 4 followed by either every 4 weeks (Q4W) (with historical radiographic evidence of joint damage) or every 8 weeks (Q8W) (without historical evidence of joint damage) dosing with the last dose at Week 52. Participants at high risk of joint damage can also be considered for Q4W dosing per investigator.
  Interventions: Drug: Guselkumab

INTERVENTIONS:
Drug: Ustekinumab — Ustekinumab will be administered as subcutaneous injection.
  Other Names: CNTO1275; STELARA
  Arms: Cohort 1: Ustekinumab
Drug: Guselkumab — Guselkumab will be administered as subcutaneous injection.
  Other Names: CNTO1959; TREMFYA
  Arms: Cohort 2: Guselkumab

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (PK), efficacy, safety and immunogenicity of ustekinumab and guselkumab in active juvenile psoriatic arthritis (jPsA).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of juvenile psoriatic arthritis (jPsA) by Vancouver criteria with exclusion of enthesitis-related arthritis (ERA). Diagnosis made >=3 months (that is, 90 days) prior to screening
* Active disease in at least greater than or equal to (>=) 3 joints at screening and at week 0 (defined as swelling or loss of motion with pain and/or tenderness. Swelling alone meets the criteria for an active arthritic joint. In the absence of swelling, loss of motion with pain or tenderness or both pain and tenderness meet the criteria for an active arthritic joint
* Have active disease despite previous non-biologic disease modifying anti-rheumatic drug (DMARD) and/or non-steroidal anti-inflammatory drug (NSAID) therapy: Non-biologic DMARD therapy is defined as taking a non-biologic DMARD for at least 12 weeks or evidence of intolerance; NSAID therapy is defined as taking an NSAID for at least 4 weeks or evidence of intolerance
* Concurrent use of methotrexate, sulfasalazine, leflunomide, oral corticosteroids or NSAIDs is permitted but must be on stable dose
* Participants must be up to date with all immunizations in agreement with current local immunization guidelines for immunosuppressed patients
* Prior use of anti-TNFα agents, IL-17 inhibitors and other biologics (except non-responders to IL-23 inhibitors) and JAK inhibitors are permitted with sufficient washout period

Exclusion Criteria:

* Participants with enthesitis-related arthritis (ERA)
* Have a history of latent or active granulomatous infection, including tuberculosis (TB), histoplasmosis, or coccidioidomycosis prior to screening
* Have a history of, or ongoing, chronic or recurrent infectious disease
* Has evidence of herpes zoster infection within 8 weeks prior to Week 0
* Have a known history of hepatitis C infection or test positive at screening

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2022-08-30 (Actual); Primary Completion 2026-12-10 (Estimated); Study Completion 2027-08-09 (Estimated)

PRIMARY OUTCOMES:
Cohort 1: Steady-state Trough Serum Concentration of Ustekinumab at Week 28 by Baseline Age Groups | Week 28
  Steady-state trough serum concentration of ustekinumab at Week 28 by baseline age groups will be reported.
Cohort 2: Steady-state Trough Serum Concentration of Guselkumab at Week 28 by Baseline Age Groups | Week 28
  Steady-state trough serum concentration of guselkumab at Week 28 by baseline age groups will be reported.
Cohort 1: Area Under the Curve at Steady-state (AUCss) Over a 12-Week Dosing Interval of Ustekinumab at Week 28 by Baseline Age Groups | Week 28
  AUCss is defined as area under the curve at steady-state over a 12-week dosing interval of ustekinumab at Week 28 by baseline age groups.
Cohort 2: AUCss Over a Dosing Interval (4 or 8 Weeks) of Guselkumab at Week 28 by Baseline Age Groups | Week 28
  AUCss is defined as area under the curve at steady-state over a dosing interval (4 or 8 weeks) of guselkumab at Week 28 by baseline age groups.
Cohort 1: Percentage of Participants with Juvenile Psoriatic Arthritis (jPsA) Achieving American College of Rheumatology (ACR) Pediatric 30 Response at Week 24 | Week 24
  Percentage of Participants with jPsA achieving ACR pediatric 30 response at Week 24 will be reported. The ACR pediatric 30 response criteria is defined as a 30 percent (%) improvement (that is, a decrease in score) from baseline in greater than or equal to (>=) 3 of the following 6 components, with worsening of >=30% in no more than 1 of the following components: physician global assessment (PGA) of disease activity, patient/participant assessment of overall well-being, number of active joints (defined as swelling or loss of motion with pain and/or tenderness), number of joints with limited range of motion, physician function by childhood health assessment questionnaire (CHAQ) and C-reactive protein (CRP).
Cohort 2: Percentage of Participants with jPsA Achieving ACR Pediatric 30 Response at Week 24 | Week 24
  Percentage of Participants with jPsA achieving ACR pediatric 30 response at Week 24 will be reported. The ACR pediatric 30 response criteria is defined as a 30% improvement (that is, a decrease in score) from baseline in >=3 of the following 6 components, with worsening of >=30% in no more than 1 of the following components: PGA of disease activity, patient/participant assessment of overall well-being, number of active joints (defined as swelling or loss of motion with pain and/or tenderness), number of joints with limited range of motion, physician function by CHAQ and CRP.

SECONDARY OUTCOMES:
Cohorts 1: Steady-state Trough Serum Concentration of Ustekinumab at Week 52 by Baseline Age Groups | Week 52
  Steady-state trough serum concentration of ustekinumab at Week 52 by baseline age groups will be reported.
Cohorts 2: Steady-state Trough Serum Concentration of Guselkumabat at Week 52 by Baseline Age Groups | Week 52
  Steady-state trough serum concentration of guselkumab at Week 52 by baseline age groups will be reported.
Cohort 1: AUCss Over a 12-Week Dosing Interval of Ustekinumab at Week 52 by Baseline Age Groups | Week 52
  AUCss is defined as area under the curve at steady-state over a 12-week dosing interval of ustekinumab at Week 52 by baseline age groups.
Cohort 2: AUCss Over a Dosing Interval (4 or 8 Weeks) of Guselkumab at Week 52 by Baseline Age Groups | Week 52
  AUCss is defined as area under the curve at steady-state over a dosing interval (4 or 8 weeks) of guselkumab at Week 52 by baseline age groups.
Cohorts 1 and 2: Percentage of Participants Achieving ACR Pediatric 30 Response at Weeks 4, 8, 12, 16, and 52 | Weeks 4, 8, 12, 16 and 52
  The ACR pediatric 30 response criteria is defined as a 30% improvement (that is, a decrease in score) from baseline in >=3 of the following 6 components, with worsening of >=30% in no more than 1 of the following components: PGA of disease activity, patient/participant assessment of overall well-being, number of active joints (defined as swelling or loss of motion with pain and/or tenderness), number of joints with limited range of motion, physician function by CHAQ and CRP.
Cohorts 1 and 2: Percentage of Participants Achieving ACR Pediatric 50 and 70 Responses at Weeks 4, 8, 12, 16, 24, and 52 | Weeks 4, 8, 12, 16, 24, and 52
  The ACR pediatric 50 and 70 responses are defined as a 50% improvement or 70% improvement (that is, a decrease in score) from baseline in >=3 of the following 6 components, with worsening of >=30% in no more than 1 of the following components: 1 of the following components: PGA of disease activity, patient/participant assessment of overall well-being, number of active joints (defined as swelling or loss of motion with pain and/or tenderness), number of joints with limited range of motion, physician function by CHAQ and CRP.
Cohorts 1 and 2: Time to Response Measured as Time to Achieving ACR Pediatric 30 | Baseline, up to Week 24
  Time to response measured as time to achieving ACR pediatric 30 will be reported.
Cohorts 1 and 2: Change from Baseline in Clinical Juvenile Arthritis Disease Activity Score (cJADAS) 10 at Weeks 4, 8, 12, 16, 24, and 52 | Baseline, up to Weeks 4, 8, 12, 16, 24, and 52
  Change from baseline in cJADAS 10 at Weeks 4, 8, 12, 16, 24, and 52 will be reported. The cJADAS is calculated as the sum of the scores of its 3 components: (1) physician global rating of overall disease activity, measured on a 10-cm horizontal visual analog scale; (2) parent/child ratings of well-being, assessed on a 10 cm horizontal line VAS; (3) number of active joints, assessed in 10 joints, for a total score ranging from 0 to 30 where 0=no activity and 30=maximum activity.
Cohorts 1 and 2: Change from Baseline in Juvenile Arthritis Disease Activity Score (JADAS) 10, 27 and 71 at Weeks 4, 8, 12, 16, 24, and 52 | Baseline, up to Weeks 4, 8, 12, 16, 24, and 52
  Change from baseline in JADAS 10, 27 and 71 at Weeks 4, 8, 12, 16, 24, and 52 will be reported. The JADAS is calculated as the sum of the scores of its 4 components: (1) physician global rating of overall disease activity, measured on a 10-cm horizontal visual analog scale; (2) parent/child ratings of well-being, assessed on a 10 cm horizontal line VAS; (3) number of active joints, assessed in 71, 27, or 10 joints (for JADAS 71, JADAS 27, and JADAS 10, respectively); (4) CRP (truncated to 0-10 mg/dL).
Cohorts 1 and 2: Change from Baseline in Psoriasis Area Severity Index (PASI) Score at Week 24 | Baseline and Week 24
  Change from baseline in PASI score at Week 24 among the participants with greater than or equal to (>=) 3% body surface area (BSA) psoriatic involvement and a PGA psoriasis score of >=2 (mild) at baseline will be reported. The PASI includes assessments of 4 areas of the body: the head and neck, the arms, the trunk, and the legs. The percentage of skin in each area affected by psoriasis is given a numeric score representing the proportion involved. The severity of the 3 plaque signs of erythema, thickness/induration, and desquamation/scaling, is assessed on a 5-point scale. The total PASI score is from 0-72, where 0=no disease and 72=more disease.
Cohorts 1 and 2: Percentage of Participants with Adverse Events (AEs) | Up to Week 68
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Cohorts 1 and 2: Percentage of Participants with Serious Adverse Events (SAEs) | Up to Week 68
  A SAE is any untoward medical occurrence that at any dose results in any of the following outcomes: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly/birth defect; suspected transmission of any infectious agent via a medicinal product or medically important.
Cohorts 1 and 2: Percentage of Participants with Reasonably Related AEs | Up to Week 68
  Percentage of participants with reasonably related AEs (including injection-site reactions and infections) will be reported.
Cohorts 1: Number of Participants with Antibodies to Ustekinumab | Weeks 52 and 68
  Number of participants with antibodies to ustekinumab (including peak titers) will be reported.
Cohorts 2 : Number of Participants with Antibodies to Guselkumab | Weeks 52 and 68
  Number of participants with antibodies to guselkumab (including peak titers) will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (50):
- United States (9):
  - Childrens Hospital Los Angeles, Los Angeles, California
  - UCLA, Los Angeles, California
  - Harvard Medical School - Boston Children's Hospital, Boston, Massachusetts
  - Northwell Health, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Legacy Emanuel Medical Center, Portland, Oregon
  - University of Utah, Salt Lake City, Utah
- Argentina (5):
  - STAT Research S A, Ciudad Autonoma Buenos Aires
  - Hospital de Ninos de Cordoba, Córdoba
  - Instituto Medico Platense, La Plata
  - Instituto Caici, Rosario
  - Centro Medico Privado de Reumatologia, San Miguel de Tucumán
- Denmark (2):
  - Aarhus Universitetshospital, Aarhus
  - Odense Universitets Hospital, Odense
- France (5):
  - CHU de Caen, Caen
  - Hopital de Bicetre, Le Kremlin-Bicêtre
  - Hopital Nord Marseille, Marseille
  - CHU de Toulouse Hopital des Enfants, Toulouse
  - Hôpital D'Enfants, Vandœuvre-lès-Nancy
- Germany (3):
  - Charite Universitatsmedizin Berlin Campus Virchow Klinikum, Berlin
  - Schon Klinik Hamburg Eilbek, Hamburg
  - Asklepios Klinik Sankt Augustin, Sankt Augustin
- Italy (5):
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia Presidio Spedali Civili, Brescia
  - Istituto Giannina Gaslini, Genova
  - Centro Specialistico Ortopedico Traumatologico Gaetano Pini CTO, Milan
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - IRCCS Ospedale Pediatrico Bambino Gesu, Roma
- Poland (3):
  - CSK, Uniwersyteckie Centrum Pediatrii im.M.Konopnickiej, Lodz
  - Centrum Zdrowia Dziecka i Rodziny im Jana Pawla II w Sosnowcu Sp z o o, Sosnowiec
  - Narodowy Instytut Geriatrii Reumatologii i Rehabilitacji im prof dr hab med Eleonory Reicher, Warsaw
- Spain (6):
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp. de La Santa Creu I Sant Pau, Barcelona
  - Hosp Reina Sofia, Córdoba
  - Hosp. Clinico Univ. de Santiago, Santiago de Compostela
  - Hosp. Infanta Luisa, Seville
  - Hosp. Univ. I Politecni La Fe, Valencia
- Turkey (Türkiye) (4):
  - Hacettepe Universitesi Hastanesi, Ankara
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul
  - Umraniye Training and Research Hospital, Istanbul
  - Kocaeli University Medical Faculty, Kocaeli
- United Kingdom (8):
  - Great Ormond Street Hospital, London
  - Royal Manchester Children's Hospital, Manchester
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Sheffield Children's Hospital, Sheffield
  - Southampton General Hospital, Southampton
  - Haywood Hospital, Staffordshire
  - Royal Stoke University Hospital, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency